CLINICAL TRIAL: NCT03773874
Title: Assessment of Analgesia, Sedation, Physical Restraints and Delirium in Patients Admitted to Spanish Intensive Care Units. ASCyD Project
Brief Title: Assessment of Analgesia, Sedation, Physical Restraints and Delirium in Spanish Intensive Care Units
Acronym: ASCyD
Status: Completed | Type: Observational
Sponsor: Hospital Universitario Getafe (Other)
Responsible Party: Principal Investigator, Susana Arias Rivera, Principal Investigator, Hospital Universitario Getafe
Other Study IDs: PY 17/22
Record Dates: First submitted 2018-10-09; First posted 2018-12-12 (Actual); Last update posted 2018-12-12 (Actual); Status verified 2018-02

CONDITIONS: Pain; Sedation; Agitation; Delirium; Restraint, Physical; Critical Care; Nursing Assessment
MeSH Terms: conditions — Pain; Psychomotor Agitation; Delirium | interventions — Restraint, Physical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Assessment — Evaluation
  Other Names: audit

SUMMARY:
This study assess which Spanish intensive care units evaluate and record, in a standardized way, levels of pain, sedation / agitation, use of physical restraints and prevalence of delirium. Also determine the use of validated assessment tools and explore levels of pain and sedation / agitation, use of physical restraints and prevalence of delirium.

DETAILED DESCRIPTION:
An observational, descriptive, cross-sectional, prospective and multicenter study was conducted to know the usual practice (audit) in critical care units and about the assessment of pain, sedation, delirium and the use of mechanical restraints.

At the same time, the level of pain, sedation / agitation and presence of delirium were evaluated in all adult patients who were admitted to the participating units with a minimum stay of 24 hours in the unit.

Process In order to obtain the largest representation of Spanish Intensive Care Units, a network of research nurses was created with coordinators in each autonomous community. The function of the coordinators was to contact and recruit units of adult critical patients within their community. Each coordinator contacted the centers (public and private), creating a network of collaborating nurses from those units who expressed their willingness to participate and who obtained the authorization of their Research Ethics Committee. Each unit was asked to contact a collaborating nurse for the project.

Once the national network of collaborating nurses was created, through the community coordinators, each password was given to each nurse to access the platform created for data entry. The platform offered access to all the documents (methodology, timeline, recommended assessment tools, navigation tutorial for the platform).

Data collection The tool used was an ad hoc survey with online access which consisted of 2 blocks. The first block asked about the characteristics of the units, the nurse-patient ratio, the existence of protocols and the usual practice for the control of pain, sedation / agitation, delirium and the use of mechanical restraints in the unit.

In the second block, questions were asked about aspects of direct assistance to patients, and direct evaluation of pain level, sedation / agitation of patients as well as the presence of delirium and mechanical containment.

Evaluation of patients included The data collection was done by direct observation and in the same period in all participating units. These data were entered into the platform through a "Patient Code", created automatically by the system.

To assess pain in patients, the investigators used two scales, for patients with the ability to communicate, the Visual Analogue Scale (VAS) scale was recommended and for patients without the ability to communicate the Scale of Behavioral Indicators of Pain (ESCID). The evaluation of the level of sedation / agitation was recommended to be carried out with the Richmond Agitation Sedation Scale (RASS) and delirium with the Confusion Assessment Method for the Intensive Care Unit (CAM-ICU).

The data on the use of tools to assess pain, sedation / agitation and delirium, as well as the recording of the use of mechanical restraints, were collected retrospectively on the nursing records of the patients evaluated, the day after their assessment.

Statistic analysis First, a descriptive analysis was made of the general characteristics of the participating units and the study population, presenting the data with means and standard deviations (SD) or medians and interquartile ranges (RIC), as appropriate. Group comparison was performed with the Student t test for quantitative variables or nonparametric tests, as appropriate, and Fischer's test or chi-square for qualitative variables. The data was analyzed with the statistical package IBM SPSS Statistics 21.0 for Windows

ELIGIBILITY:
Inclusion Criteria:

* All adult patients who were admitted to the participating units at the time of the audit and had a minimum stay of 24 hours in the unit.

Exclusion Criteria:

* no criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients who were admitted to the participating units at the time of the audit and had a minimum stay of 24 hours in the unit.
Sampling Method: Non-Probability Sample
Enrollment: 1574 (Actual)
Dates: Start 2018-02-12 (Actual); Primary Completion 2018-02-25 (Actual); Study Completion 2018-03-11 (Actual)

PRIMARY OUTCOMES:
Communicative patient's pain with Numeric Rating Scale (NRS) in critical care units. | one day
  Primary assessment of pain. NRS scale's range from 0 to 10. 0: no pain; 1-3: light pain; 4-6: moderate pain; 7-10: severe pain
"Non communicative" patient's pain with Behavioural Indicators of Pain Scale (ESCID) in critical care units. | one day
  Primary assessment of pain ESCID scale's range from 0 to 10. 0: no pain; 1-3: light pain; 4-6: moderate pain; 7-10: severe pain
Communicative and "no communicative" patient's sedation/agitation level's with Richmond Agitation Sedation Scale (RASS) in critcal care units. | one day
  Primary assessment of sedation/agitation level' s. RASS scale range from -5 to +5. -4 to -5: depth sedation; -3 to -1: light sedation; 0: aware; +1 to +4: agitation.
Communicative and "no communicative" patient's delirium prevalence with Confusion Assessment Method for the Intensive Care Unit (CAM-ICU) in critical care units | one day
  Primary assessment of delirium
Use of physical restraints on Communicative and "no communicative" patient's in critical care units | one day
  Primary assessment of use of physical restraints

SECONDARY OUTCOMES:
use of validated scale of pain: Numeric Rating Scale (NRS) | one day
  use of validated scales of pain for communicative patients. NRS scale's range from 0 to 10. 0: no pain; 1-3: light pain; 4-6: moderate pain; 7-10: severe pain.
use of validated scale of pain: Visual Analog Scale (VAS) | one day
  use of validated scales of pain for communicative patients. VAS, scale's range from 0 to 10. 0: no pain; 1-3: light pain; 4-6: moderate pain; 7-10: severe pain.
use of validated scale of pain: Campbell scale | one day
  use of validated scales of pain for "non communicative" patients. Campbell scale's range from 0 to 10. 0: no pain; 1-3: light pain; 4-6: moderate pain; 7-10: severe pain.
use of validated scale of pain: Behavioural Indicators of Pain Scale (ESCID) | one day
  use of validated scales of pain for "non communicative" patients. ESCID scale's range from 0 to 10. 0: no pain; 1-3: light pain; 4-6: moderate pain; 7-10: severe pain.
use of validated scales of pain: Behavioral Pain Scale (BPS) | one day
  use of validated scales of pain for "non communicative" patients. scale's range from 3 to 12; 3: no pain, high number more pain.
use of validated scales of pain: Critical-Care Pain Observation Tool (CPOT) | one day
  use of validated scales of pain for "non communicative" patients. CPOT: range from 0 to 8; 0-2: no pain, > 2 pain.
use of validated scales of sedation/agitation (RASS) | one day
  use of validated scales of sedation/agitation patients. RASS scale range from -5 to +5. -4 to -5: depth sedation; -3 to -1: light sedation; 0: aware; +1 to +4: agitation.
use of validated scales of sedation/agitation (Ramsay scale) | one day
  use of validated scales of sedation/agitation patients. Ramsay score from 1 to 6; 1: anxious, agitated restless, 2: cooperative, oriented, tranquil, 3: responsive to commands only, 4: brisk response to light glabellar tap or loud auditory stimulus, 5: sluggish response to light glabellar tap or loud auditory stimulus, 6: no response to light glabellar tap or loud auditory stimulus.
use of validated scales of delirium (Intensive Care Delirium Screening Checklist (ICDSC)) | one day
  Use of validated scales of delirium. ICDSC is positive (delirium present) or negative (no delirium).
use of validated scales of delirium (CAM-ICU) | one day
  Use of validated scales of delirium. CAM-ICU is positive (delirium present) or negative (no delirium).
protocols of pain and sedation | one day
  Presence of protocols in the critical care units
protocols of use of physical restraints | one day
  Presence of protocols in the critical care units
protocols of management of delirium | one day
  Presence of protocols in the critical care units

CONTACTS AND LOCATIONS:
Overall Officials: Susana Arias-Rivera, RN, Principal Investigator — Hospital Universitario de Getafe
Locations (1):
- Hospital Universitario de Getafe, Getafe, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Arias-Rivera S, Lopez-Lopez C, Frade-Mera MJ, Via-Clavero G, Rodriguez-Mondejar JJ, Sanchez-Sanchez MM, Acevedo-Nuevo M, Gil-Castillejos D, Robleda G, Cachon-Perez M, Latorre-Marco I; Equipo ASCyD. Assessment of analgesia, sedation, physical restraint and delirium in patients admitted to Spanish intensive care units. Proyecto ASCyD. Enferm Intensiva (Engl Ed). 2020 Jan-Mar;31(1):3-18. doi: 10.1016/j.enfi.2018.11.002. Epub 2019 Apr 16. English, Spanish. PMID 31003871